CLINICAL TRIAL: NCT04248192
Title: A Study to Evaluate the Safety, Immunologic, and Virologic RESponses of Donor Derived (DD) HIV-Specific T-cells (HST) With Non-escaped Epitope Targeting (NEETs) in HIV-Infected Individuals on Antiretroviral Therapy Following Allogeneic Bone Marrow Transplantation (alloRESIST)
Brief Title: Evaluate the Safety, Immunologic, and Virologic Responses of Donor Derived (DD) HIV-Specific T-cells (HST) in HIV-infected Individuals Following Allogeneic Bone Marrow Transplantation (alloRESIST)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director, Center for Cancer and Immunology Research, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012451
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: HIV-Infected Individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Donor Derived HIV-Specific T-cells (DD HST-NEETs) (Experimental): Participants who meet specified inclusion criteria including neutrophil recovery post-transplant and for whom donor products have passed release testing will receive DD HST-NEETs at a dose of 2x107/m2 within 30 days of screening visit.
  Interventions: Biological: DD HST-NEETs

INTERVENTIONS:
Biological: DD HST-NEETs — HIV-infected individuals following Allogeneic Bone Marrow Transplantation (alloBMT) will be treated with DD HST-NEETS therapy. Participants and donors will be screened for eligibility. Eligible donors will undergo a blood draw of up to 300mL to allow production of allogeneic DD HST-NEETs. Participants, who meet specified inclusion criteria including neutrophil recovery post-transplant and for whom donor products have passed release testing, will receive DD HST-NEETs at a dose of 2x107/m2 within 30 days of screening visit.

SUMMARY:
This is a multi-site phase 1 study of the safety, immunologic and virologic responses of ex vivo expanded donor-derived (DD) HIV-1 multi-antigen specific T-cell (HST) with non-escaped epitope targeting (NEET) therapy as a therapeutic strategy in HIV-infected individuals following Allogeneic Bone Marrow Transplantation (alloBMT).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety of donor-derived allogeneic expanded HIV-specific T-cell therapy (DD HST-NEETs) in HIV-infected alloBMT recipients on ART. Eligible donors will undergo a blood draw of up to 300mL to allow production of allogeneic DD HST-NEETs. Participants who meet specified inclusion criteria including neutrophil recovery post-transplant and for whom donor products have passed release testing will receive DD HST-NEETs at a dose of 2x107/m2 within 30 days of screening visit.

ELIGIBILITY:
Inclusion Criteria:

Participant Inclusion Criteria at Screening:

* Age ≥18 years.
* Confirmation of HIV-1 infection. Any licensed ELISA test kit which is confirmed by Western blot or Multispot HIV-1/HIV-2 assay prior to screening. HIV culture, HIV antigen, plasma HIV RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
* On effective antiretroviral therapy.
* Ability and willingness of participant to continue and be compliant with ART throughout the study.
* Hematologic malignancy that qualifies for standard of care alloBMT according to JHU criteria.
* Potential participant must have adequate organ function for standard of care alloBMT according to JHU criteria.
* No active HCV infection. (If seropositive, participant must have no measureable HCV RNA within 30 days of enrollment).
* No active HBV infection (If seropositive, participant must have no measureable HBV DNA or HBsAg+ within 30 days of enrollment).
* Ability and willingness of participant to give written informed consent.
* Ability and willingness to communicate effectively with study personnel; considered reliable, willing, and cooperative in terms of compliance with the Protocol requirements.
* Ability and willingness to provide adequate locator information and contact information for at least 2 adults who can reach the participant within 24 hours

Participant Inclusion Criteria for DD HST-NEETs Infusion:

* Karnofsky score of ≥ 70.
* ANC ≥ 250/µL.
* Bilirubin ≤ 2x upper limit normal or direct bilirubin normal.
* AST ≤ 3x upper limit normal.
* Serum creatinine ≤ 2x upper limit normal.
* Hgb ≥ 7.0 g/dL.
* Pulse oximetry of > 90% on room air.
* Negative pregnancy test in female participants if applicable (childbearing potential).
* Written informed consent signed by participant or guardian.
* Steroids less or equal to 0.5 mg/kg/day prednisone.

Donor Inclusion Criteria for Procurement for DD HST-NEETS Manufacturing:

* Donors for allogeneic (i.e. HLA matched or mismatched related or unrelated) hematopoietic cell transplants who have fulfilled eligibility for and consented to stem cell donation as per JHU standard operating procedures.
* Donor must be in good health based on institutional guidelines.
* Female donors of childbearing age must have a negative pregnancy test and must not be lactating.
* It is understood that medical clearance from the donor will be sought within the timeline per the National Marrow Donor Program (NMDP) rules.
* The hematopoietic cell donor will have already been selected by the JHU BMT Donor Selection Committee.
* Donor or parent/guardian capable of providing informed consent

Exclusion Criteria:

Participant Exclusion Criteria DD HST-NEETs Infusion:

* Participants receiving ATG, or Campath or other immunosuppressive T-cell monoclonal antibodies within 28 days.
* Participants with uncontrolled infections. For bacterial infections, participants must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections participants must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection.
* Participants who have received donor lymphocyte infusion (DLI) within 28 days.
* Active and uncontrolled relapse of malignancy.
* Participants with active acute GVHD grades II-IV
* Participants with bronchiolitis obliterans syndrome or serositis
* Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, pneumococcal polysaccharide) within 28 days prior to study entry.
* Inability to comply with study requirements, which could impact study integrity and/or safety.

Donor Exclusion Criteria for Procurement for DD HST-NEETs Manufacturing:

• Donor exclusion criteria will be followed as per institution standard operating procedures (SOPs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Any ≥ Grade 3 Adverse Events (as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0) | 45 days
  Any ≥ Grade 3 Adverse Events will be measured by number of participants who experience Dose Limiting Toxicity which is attributable to the DD HST-NEETS administration.

SECONDARY OUTCOMES:
The feasibility of manufacturing of DD HST-NEETs | 3 years
  Feasibility of the manufacturing process will be measured by generation of the cells in 4 or more donors (i.e., a rate of 50% of more).
The HIV reservoir measurements | 3 years
  Summarize the HIV reservoir measurements over the pre-BMT, pre-DD HST-NEETs infusion, post-infusion period to assess any change in the HIV reservoir following infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ambinder, MD, PhD, Principal Investigator — Johns Hopkins University; Michael Keller, MD, Principal Investigator — CNMC
Locations (1):
- Johns Hopkins University(Jhu), Baltimore, Maryland, United States